CLINICAL TRIAL: NCT02149147
Title: Variety of Physical Activity in Normal to Overweight Adults Who Are Regularly Active
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Other Study IDs: 9492 B
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Overweight
Keywords: physical activity; environmental factors; variety; MVPA
MeSH Terms: conditions — Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical Activity Variety: participants will complete the Self-Efficacy questionnaire, the Physical Activity Enjoyment Scale, the Behavioral Regulation in Exercise-2 questionnaire, and an Outcome Expectations questionnaire. Participants will be instructed to wear the SenseWear® armband which will measure physical activity-related energy expenditure for the course of the study. The armband will be worn every day for at least 10 hours per day. In addition, participants will be asked to complete a physical activity diary to record their physical activity as well as additional information about the environment in which the physical activity was conducted. Participants will be instructed to engage in their normal physical activity regimen, wear the armband, and complete the physical activity diary for 3 weeks.

SUMMARY:
The purpose of this study is to investigate the variety of physical activity, a cross-sectional design will be used. The data collected will provide descriptive details about how people are engaging in physical activity, as well details about the environment they are in while engaging in physical activity.

DETAILED DESCRIPTION:
Many individuals, particularly those who are obese, are inactive and increasing physical activity continues to be a challenge, thus, developing strategies that assist individuals in engaging and sustaining high levels of physical activity is imperative.1,2 Incorporating a variety of activities into a physical activity program is a strategy that may be promising for increasing physical activity levels.3 Data from the National Health and Nutrition Examination Survey (NHANES) showed that individuals who reported engaging in a variety of activities (i.e., walking + other leisure-time activities) were more likely to meet national physical activity recommendations compared to those who reported no variety (i.e., only walking).4 In another study, the investigators found that overweight participants in an 18-month behavioral lifestyle intervention who reported physical activity variety (i.e., ≥ 2 activities) at 6 months had higher self-reported physical activity-related energy expenditure and a lower body mass index (BMI) at 18 months than those who reported no physical activity variety (i.e., only 1 activity).5 Additionally, the investigators have also found that performing a variety of activities is related to greater engagement in objectively measured moderate- to vigorous-intensity physical activity in both successful weight loss maintainers and normal weight individuals.6 Based on the literature available, it appears that increasing the number of activities in a physical activity regimen can assist with increasing engagement of physical activity. However, physical activity variety has primarily been examined by summing the number of different activities a person engages in (i.e., walking + other leisure-time activities). Other environmental factors, including location, visual and auditory stimuli, and the number and types of people engaging in physical activity in close proximity, may impact on the degree of variety of differing physical activities that people engage in. Thus, the purpose of this study is to collect more information about physical activity variety.

Specific Aims:

Specific Aim 1. To determine the average minutes of moderate- to vigorous-intensity physical activity participants engage in.

Specific Aim 2. To determine if environmental factors influence the degree of variety of physical activities that participants engage in.

Specific Aim 3. To determine if the average number of minutes of moderate- to vigorous-intensity physical activity increases as the variety of physical activities increases.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 29.9 kg/m2.

Exclusion Criteria:

* Have a metal allergy (which would prevent the ability of a participant to wear the SenseWear® armband from BodyMedia® used in the proposed study).
* Self-report engaging in less than 30 minutes/week of moderate- to vigorous-intensity physical activity over the previous week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be 50 men and women, recruited from flyers posted on the University of Tennessee-Knoxville campus and in local gyms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Baseline, 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee-Knoxville
Locations (1):
- University of Tennessee-Knoxville: Jesse Harris Building, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this program is being conducted — http://nutrition.utk.edu/healthy-eating-and-activity-laboratory/